CLINICAL TRIAL: NCT04891692
Title: Effect of Neuromuscular Electrical Stimulation Using the StimaWELL 120MTRS System on Multifidus Muscle Morphology and Function in Patients With Chronic Low Back Pain
Brief Title: Effect of Neuromuscular Electrical Stimulation in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCER 20-21-07
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-08

CONDITIONS: Low Back Pain; Paraspinal Muscles
Keywords: Diagnostic Imaging; Electrical Stimulation Therapy; Low Back Pain; Paraspinal Muscles
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phasic Treatment Group (Experimental): Muscle therapy for the lumbar spine at the StimaWell 120MTRS system's phasic setting. Treatment at 3 kHz, modulation 50 Hz. Supervised 10 week intervention, 2 times a week. Treatment time of 20 minutes for the first 3 weeks, 25 minutes for the second 3 weeks, and 30 minutes for the final 4 weeks. 120MTRS system recalibration every fifth treatment.
  Interventions: Device: StimaWell 120MTRS system
- Combined Treatment Group (Experimental): Muscle therapy for the lumbar spine at the StimaWell 120MTRS system's combined (tonic and phasic) setting. Treatment at 3 kHz, modulation 4 Hz and 50 Hz. Supervised 10 week intervention, 2 times a week. Treatment time of 20 minutes for the first 3 weeks, 25 minutes for the second 3 weeks, and 30 minutes for the final 4 weeks. 120MTRS system recalibration every fifth treatment.
  Interventions: Device: StimaWell 120MTRS system

INTERVENTIONS:
Device: StimaWell 120MTRS system — Medium-frequency electrotherapy device that delivers current via up to 12 channels. The device also provides heat therapy up to 40°C.

SUMMARY:
This study evaluates the effect of a 10-week long intervention with the StimaWELL 120MTRS system on multifidus morphology and function in individuals with chronic low back pain. Half the participants will receive muscle therapy at the device's phasic setting, while half will receive muscle therapy at the device's combined setting. This study also evaluates the acute effect of a single treatment with the StimaWELL 120MTRS on multifidus stiffness in individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific LBP (>3 months), defined as pain in the region between the lower ribs and gluteal folds, with or without leg pain.
* Aged between 18 to 60 years old.
* English or French speakers
* At least a 4/10 score on an 11-point Numerical Pain Rating Scale (NPRS) for pain intensity.

The score will be the average of current pain, and best and worst pain over the previous week.

* At least a 'moderate' Modified Oswestry Disability Index (ODI) score.
* Able to undergo MRI exam.

Exclusion Criteria:

* Currently undergoing or having received physical therapy treatment in the previous month
* Consistent motor control training for the low back and / or consistent weightlifting, power-lifting, bodybuilding, or strongman training in the previous 6 weeks
* History of lumbar surgery
* Presence of positive lumbosacral dermatomes or myotomes
* Presence of disease which could affect the stiffness of muscle tissue (collagen tissue disease, hemiplegia, multiple sclerosis, blood clots)
* Presence of systemic disease (cancer, metabolic syndrome)
* Presence of rheumatoid arthritis
* Presence of spinal stenosis, fracture, infection, or tumor
* Presence of lumbar scoliosis greater than 10 degrees
* Presence of cardiac arrhythmia
* Pregnant and breastfeeding women
* Individuals with epilepsy
* Individuals at risk for serious bleeding
* Individuals with pacemakers or metal implants
* Individuals with aneurysms or heart valve clips
* Individuals with tattoos or piercings in the lumbar spine
* Individuals who have taken prescribed muscle relaxants more than once a week over the past month
* BMI > 30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Change in multifidus muscle size (cross-sectional area) | Baseline, after 10 weeks
  Multifidus muscle cross-sectional area measurements will be obtained from magnetic resonance imaging (MRI) at L4-L5 and L5-SI spinal levels.
Change in multifidus muscle fat infiltration | Baseline, after 10 weeks
  Multifidus muscle fatty infiltration (composition) measurements will be obtained from magnetic resonance imaging (MRI) at L4-L5 and L5-S1 spinal levels
Change in multifidus muscle function (% thickness change) | Baseline, after 10 weeks
  Multifidus muscle function, expressed as the % thickness change from a rested to contracted position via prone contralateral arm lifts will be assessed by ultrasound.
Change in multifidus muscle stiffness | Baseline, after 10 weeks
  Multifidus muscle stiffness, obtained at rest in a prone position, with prone contralateral arm lifts, and in a standing position, will be assessed by ultrasound (shear-wave elastography)
Change in multifidus muscle stiffness | Before and 15 minutes after 3rd treatment
  Multifidus muscle stiffness, obtained at rest in a prone position, and in a standing position, will be assessed by ultrasound (shear-wave elastography)

SECONDARY OUTCOMES:
Change in the Numerical Pain Rating Scale (NPRS) for low back pain intensity at present | Baseline, before and after each treatment, after 10 weeks
  The NPRS measures pain intensity on a scale of 0 - 10, with 0 being no pain, and 10 being the worst pain imaginable
Change in the Numerical Pain Rating Scale (NPRS) for low back pain intensity (best and worst pain over previous week) | Baseline, prior to 11th treatment, after 10 weeks
  The NPRS measures pain intensity on a scale of 0 - 10, with 0 being no pain, and 10 being the worst pain imaginable
Change in the Numerical Pain Rating Scale (NPRS) for low back pain intensity (sitting and with movement over past 24h) | Baseline, prior to 11th treatment, after 10 weeks
  The NPRS measures pain intensity on a scale of 0 - 10, with 0 being no pain, and 10 being the worst pain imaginable
Change in the Numerical Pain Rating Scale (NPRS) for overall leg pain intensity in the past week | Baseline, prior to 11th treatment, after 10 weeks
  The NPRS measures pain intensity on a scale of 0 - 10, with 0 being no pain, and 10 being the worst pain imaginable
Change in the Oswestry Disability Index (ODI) | Baseline, prior to 11th treatment, after 10 weeks
  The ODI is used to measure the participant's level of disability in relation to LBP. It is a 10-item scale in which each item is rated from 0-6. Higher scores indicate greater disability.
Change in the Pain Catastrophizing Scale (PCS) | Baseline, prior to 11th treatment, after 10 weeks
  The PCS is a 13-item questionnaire that assesses the participant's level of catastrophizing. Each item is rated from 0-4 for a possible total of 52. Higher scores indicate greater catastrophizing.
Change in the Brief Pain Inventory - Interference (BPI) | Baseline, prior to 11th treatment, after 10 weeks
  The BPI-I is a 7-item questionnaire that measures how pain interferes with activities of daily living. Each item is rated from 0-10. Higher scores indicative greater interference.

CONTACTS AND LOCATIONS:
Locations (1):
- PEFORM Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortin M, Wolfe D, Dover G, Boily M. The effect of phasic versus combined neuromuscular electrical stimulation using the StimaWELL 120MTRS system on multifidus muscle morphology and function in patients with chronic low back pain: a randomized controlled trial protocol. BMC Musculoskelet Disord. 2022 Jul 1;23(1):627. doi: 10.1186/s12891-022-05578-1. PMID 35773711